CLINICAL TRIAL: NCT00458315
Title: Randomized Fase II Trial: Comparing Cisplatin, Paclitaxel and Gemcitabine Versus Cisplatin, Paclitaxel, Gemcitabine and Avastin in Patients With Unknown Primary Tumors
Brief Title: Cisplatin/Paclitaxel/Gemcitabine +/- Avastin in Patients With Unknown Primary Tumor
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: never been started
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Gedske Daugaard, dr., Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cis/Gem/Tax +/- Avastin
Record Dates: First submitted 2007-04-06; First posted 2007-04-10 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2009-09

CONDITIONS: Unknown Primary Tumors
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — Cisplatin; Paclitaxel; Gemcitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cisplatin
Drug: Paclitaxel
Drug: Gemcitabine
Drug: Avastin (Bevacizumab)

SUMMARY:
The purpose of this study is to investigate the efficacy of Cisplatin, Paclitaxel, Gemcitabine +/- Avastin (Bevacizumab) in patients with unknown primary tumors.

DETAILED DESCRIPTION:
Upon determination of eligibility, all patients will be randomly assigned to one of two treatment arms:

Arm A: Cisplatin, Paclitaxel and Gemcitabine

* Cisplatin 75 mg/m2 IV infusion, Day 1
* Paclitaxel 175 mg/m2 IV infusion, Day 1
* Gemcitabine 1000 mg/m2 IV infusion, Day 1 and 8

Arm B: Cisplatin, Paclitaxel, Gemcitabine and Avastin (Bevacizumab)

* Cisplatin 75 mg/m2 IV infusion, Day 1
* Paclitaxel 175 mg/m2 IV infusion, Day 1
* Gemcitabine 1000 mg/m2 IV infusion, Day 1 and 8
* Bevacizumab 7,5 mg/m2 IV infusion, Day 1

Patients will be stratified by number of metastatic sites (one versus two or more) and the level of Lactate Dehydrogenase (normal versus high).

The regimens will be repeated every 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Unknown primary tumors
2. ECOG performance status 0-1
3. Adequate kidney, liver and bone marrow function
4. No prior chemotherapy
5. Life expectancy > 3 months

Exclusion Criteria:

1. The following specific syndromes:

   * Squamous carcinoma limited to cervical glands
   * Women with adenocarcinoma isolated to axillary nodes
   * Women with adenocarcinoma isolated to peritoneal involvements
   * Young men (<55 years) with growing mid-line tumors where a germ cell tumor could be expected
   * Neuroendocrine carcinomas
2. Tumor located close to major blood vessels and judged to possess a high risk of serious bleeding
3. Any significant cardiac disease
4. Clinically significant peripheral vascular disease
5. History of myocardial infarction or stroke within 6 months
6. Evidence of coagulopathy
7. Use of ASA, NSAIDs or clopidogrel
8. Pregnancy or breast feeding
9. Ongoing therapeutic anti-coagulation
10. Hypertension with blood pressure > 150/100 mmHg
11. Brain metastases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05; Primary Completion 2007-08 (Actual); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival
Response

SECONDARY OUTCOMES:
Toxicity
Response Duration

CONTACTS AND LOCATIONS:
Overall Officials: Gedske Daugaard, MD, Principal Investigator — Rigshospitalet, Dept of Oncology
Locations (1):
- Rigshospitalet, Dept of Oncology, Copenhagen, Denmark